CLINICAL TRIAL: NCT02485860
Title: Interest in the Use of Dressings With Honey for Wound Healing After Excision of Pilonidal Cyst
Acronym: Pilomiel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHD018-15
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Results first posted 2023-10-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Pilonidal Cysts
Keywords: pilonidal cysts; Cavity wound; long healing; honey
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard dressings (No Intervention): In general, the dressings made are either of the type :
  * Algosteril® (round or flat wick) + Mepilex® border
  * or AquacelTM ExtraTM + AquacelTM Foam
- standard dressings with sterile honey (Experimental): Melectis G
  Interventions: Device: Melectis G

INTERVENTIONS:
Device: Melectis G
  Arms: standard dressings with sterile honey

SUMMARY:
The management of pilonidal cysts is a skin excision and under deep skin. Scarring requires regular dressings (daily for 15 days and then every 48 hours) until complete healing. This healing is obtained on average in 68 days. Some patients have difficulties in healing with a final healing achieved on average in 95 days. Some teams use honey to promote wound cavitary wounds (wound infection, pressure ulcers, varicose wound). The acceleration of wound healing is due to antibacterial properties and hyperosmolarity to reduce secretions. ) The use of honey in pilonidal cysts is not evaluated and may accelerate healing.

ELIGIBILITY:
Inclusion Criteria:

* Cavity Wound to 6 weeks of a pilonidal cyst excision
* Bloodless wound
* Pilonidal cyst not recurred
* Age : 18 years and older
* Signature of informed consent
* In the capacity to understand the study

Exclusion Criteria:

* Bleeding wound
* Refused to participate in Protocol
* Patient immunocompromised
* Recurrent pilonidal cyst
* Patients on long-term corticosteroid
* Patient deprived of liberty, under guardianship
* Patient unable to understand the study
* Allergy or hypersensitivity to honey
* Allergy Or hypersensitivity to hyaluronic acid
* Allergy or hypersensitivity to guar gum
* Allergy or hypersensitivity to pectin
* Known allergy to propolis (potentially present in honey)
* Sensitivity to zinc oxide
* Sensitivity known dressings used in this trial or any component
* Diabetes Non-insulin or insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 890 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emeric ABET, PH, Principal Investigator — Centre Hospitalier Departemental Vendee
Locations (1):
- Centre Hospitalier Departemental Vendée, La Roche-sur-Yon, France

REFERENCES:
- [Result] Abet E, Jean MH, Greilsamer T, Planche L, Maurice F, Brau-Weber AG, Denimal F. The value of honey dressings in pilonidal cyst healing: a prospective randomized single-center trial. Tech Coloproctol. 2023 Sep;27(9):721-727. doi: 10.1007/s10151-022-02740-8. Epub 2023 Jan 4. PMID 36598614

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 890 enrolled participants, 100 met inclusion criteria and were randomized to treatment
Groups:
- Standard dressings: Algosteril® + Mepilex® border or AquacelTM ExtraTM + AquacelTM Foam
Period: Overall Study
Arm/Group | Standard dressings | Standard dressings with sterile honey
Started | 50 | 50
Completed | 44 | 47
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 4 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Health context (COVID-19) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Dressings: Algosteril® (round or flat wick) + Mepilex® border or AquacelTM ExtraTM + AquacelTM Foam
- Total: Total of all reporting groups
Arm/Group | Standard Dressings | Standard Dressings With Sterile Honey | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25 (8) | 24 (8) | 24 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 19 | 43
  Male | 26 | 31 | 57
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Healing Time
Time Frame: from randomization to 180 days maximum
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard dressings | Standard dressings with sterile honey
Number analyzed (Participants) | 50 | 50
Days | 78 (55) | 61 (44)
Statistical Analysis 1: Comparison: Standard dressings vs Standard dressings with sterile honey; Test type: Superiority; p = 0.094, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From inclusion to the end of follow-up (D180 or healing)
Arm/Group | Standard dressings | Standard dressings with sterile honey
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/50
Other Adverse Events (participants affected / at risk) | 20/50 | 28/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard dressings (N=50) | Standard dressings with sterile honey (N=50)
Pilonidal cyst with abscess (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard dressings (N=50) | Standard dressings with sterile honey (N=50)
Application site haemorrhage (General disorders) | 8 | 14
Wound dehiscence (Injury, poisoning and procedural complications) | 5 | 13
Application site pain (General disorders) | 4 | 9
Application site irritation (General disorders) | 1 | 3
Application site pruritus (General disorders) | 1 | 6
Impaired healing (General disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT02485860/Prot_SAP_000.pdf